CLINICAL TRIAL: NCT04109911
Title: Effect of Fermented Oyster Extract on Musculoskeletal Biomarkers in Relative Sarcopenia Adults: a Randomized, Double-blinded, Placebo-controlled Trial
Brief Title: Effect of Fermented Oyster Extract on Musculoskeletal Biomarkers in Relative Sarcopenia Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pusan National University Yangsan Hospital (Other)
Responsible Party: Principal Investigator, Sang Yeoup Lee, Professor, Pusan National University Yangsan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 02-2019-013
Record Dates: First submitted 2019-09-27; First posted 2019-10-01 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Muscular Sarcoidosis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fermented oyster extract group (Experimental): This group takes fermented oyster extract for 12 weeks
  Interventions: Dietary Supplement: Fermented oyster extract
- Placebo group (Placebo Comparator): This group takes placebo for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Fermented oyster extract — Fermented oyster extract 1,200 mg/day for 12 weeks
  Arms: Fermented oyster extract group
Dietary Supplement: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
The investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the fermented oyster extract on muscle strength, muscle mass, and muscle function in healthy adults for 12 weeks.

DETAILED DESCRIPTION:
Previous studies have indicated that fermented oyster extract may have the ability to prevent skeletal muscle atrophy. Therefore, the investigators conduct a randomized, double-blind, placebo-controlled study to investigate the effects of the fermented oyster extract on muscle strength, muscle mass, and muscle function in healthy adults; the safety of the compound are also evaluate. The Investigators examine the peak torque/body weight at 60°/s knee extension, handgrip strength, skeletal muscle mass, physical performance, and metabolic parameters at baseline, as well as after 4 and 12 weeks of intervention. Fifty-four healthy adults were administered either 1,200 mg of fermented oyster extract or a placebo each day for 12 weeks;

ELIGIBILITY:
Inclusion Criteria:

* <110% of the standard lean body mass as measured using the body composition analyzer
* Body-mass index (BMI) ranging from 18.5 to 30.0 kg/m2

Exclusion Criteria:

* Abnormal liver or renal function (i.e., serum aminotransferase activity > 60 IU/L and serum creatinine concentrations > 1.2 mg/dL)
* Diabetes (diagnosed clinically or fasting glucose level > 126 mg/dL)
* History of fracture during the previous year
* Uncontrolled hypertension
* History of serious cardiac disease such as angina or myocardial infarction
* History of gastrectomy
* History of medication for psychiatric disease
* Administration of oriental medicine including herbs within the past 4 weeks Evidence of relatively high skeletal mass (more than 110% of the standard lean body mass as measured using the body composition analyzer

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
muscle strength | 12 weeks
  the peak torque/body weight at 60°/s knee extension

CONTACTS AND LOCATIONS:
Overall Officials: Sang Yeoup Lee, MD, Principal Investigator — Pusan National University Yangsan Hospital
Locations (1):
- Pusan National University Yangsan Hospital, Yangsan, Gyeungsangnam-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee YL, Lee SY. Effect of fermented oyster (Crassostrea gigas) extracts and regular walking on muscle strength and mass in older adults with relatively low muscle mass: A randomized controlled trial. Front Nutr. 2022 Jul 25;9:935395. doi: 10.3389/fnut.2022.935395. eCollection 2022. PMID 35958254